CLINICAL TRIAL: NCT05137171
Title: A Single-center, Single-arm, Prospective Phase II Clinical Study of the Efficacy and Safety of AK105 Combined With Anlotinib in the Treatment of Persistent, Recurrent, and Metastatic Cervical Cancer
Brief Title: AK105 Combined With Anlotinib in Patients With Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Ruixia Guo, Director, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-GO-025
Record Dates: First submitted 2021-11-15; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Cervical Cancer
Keywords: AK105,anlotinib,recurrent,metastatic
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — anlotinib; penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK105 and anlortinib (Experimental): AK105 200mg iv q3w;anlotinib 12mg 2w on/1w off po qd;21 days as a cycle until PD,intolerable toxicity, investigator or patient decision to withdraw, non-adherence to treatment or trial procedures.
  Interventions: Drug: AK105 and anlotinib

INTERVENTIONS:
Drug: AK105 and anlotinib — AK105(penpulimab): 200mg, every 3 weeks, 21 days as a treatment cycle;Anlotinib: 12mg, 2 weeks on/1 week off, 21 days as a treatment cycle;Treatment will continue until confirmed radiographic progression,unacceptable toxicity, investigator or patient decision to withdraw, non-adherence to treatment or trial procedures.
  Other Names: penpulimab and anlotinib

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of AK105 (anti-PD-1 mab) combined with Anlotinib Hydrochloride in the treatment of persistent, recurrent and metastatic cervical cancer.

DETAILED DESCRIPTION:
Patients with persistent,recurrent or metastatic cervical cancer (histologic types include squamous cell carcinoma, adenocarcinoma, and adenosquamous carcinoma) who had received at least once platinum-based systemic chemotherapy were enrolled.Eligible patients receive AK105 200 mg by intravenous (iv.) infusion every 3 weeks (Q3W),and anlotinib 12mg 2 weeks on/1 week off orally(Q3W).Imaging will be performed after the 3th AK105 administration as 3 cycles.This study is an open,single-arm,single-center clinical trial,and all the patients will receive AK105 and anlotinib treatment until radiographic progression,unacceptable toxicity, investigator or patient decision to withdraw, non-adherence to treatment or trial procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participated in the study and signed informed consent;
2. Age between 18 and 75;
3. Agreed to detect the expression status of PD-L1 biomarker;
4. ECOG score is 0 or 1, and the expected survival time is not less than 3 months;
5. Histologically confirmed recurrent or metastatic squamous cell carcinoma, adenocarcinoma, and adenosquamous carcinoma with documented disease progression. Note that histological confirmation of the original primary tumor is required by pathological reports;
6. Patients with recurrent or metastatic cervical cancer who had received at least once platinum-based systemic chemotherapy were included;
7. The patient is not suitable for local treatment (surgery or radiotherapy cannot be performed);
8. Patients with measurable lesions as defined in RECIST1.1 criteria;
9. The main organs function is well, and the laboratory test indexes meet the following requirements:(1) Routine blood test (no blood transfusion or hematopoietic stimulating factor was used within 7 days before screening) :① Hemoglobin (HB) ≥ 90g/L;② Absolute neutrophil count (ANC) ≥1.5×109/L;③ Platelet (PLT) ≥ 80×109/L;(2) Blood biochemical test (no blood transfusion or albumin within 7 days before screening) :① ALT and AST ≤2.5 × ULN (liver/bone metastasis ≤5 × ULN;Bone metastases ≤5 ULN);② Serum total bilirubin (TBIL) ≤1.5 × ULN;③ Serum Cr≤1.5×ULN or creatinine clearance ≥60 mL /min;(3) Coagulation function test:① Activated partial thrombin time (APTT), international standardized ratio (INR), prothrombin time (PT) ≤ 1.5×ULN;② Doppler ultrasound assessment: left ventricular ejection fraction (LVE F)≥ 50%;
10. Any toxic side effects of previous chemotherapy have been recovered to ≤CTCAE1 or baseline level;
11. The patient has the ability to take medication orally;
12. Women of reproductive age must agree to use a highly effective method of contraception during the study period and for 6 months after the last administration of the study drug;Negative serum or urine pregnancy test within 7 days prior to study enrollment and must be non-lactating subjects;

Exclusion Criteria:

1. Patients with a history or signs of brain metastases;
2. Prior use of bevacizumab, antiangiogenic drugs and other antiangiogenic drugs;
3. Received anti-tumor monoclonal antibody treatment within 4 weeks before enrollment; Had previously received other PD-1/PD-L1 antibodies and anti-CTLA-4 (cytotoxic T-lymphocyte associated antigen-4) therapy.
4. Patients were receiving immunosuppressant or systemic hormone therapy for immunosuppression (dose > 10mg/ day of prednisone or other equivalent hormone) and were still using 2 weeks prior to enrollment
5. Participate in other clinical trials or complete other clinical trials within 4 weeks;
6. Abnormal coagulation function (INR > 2.0, PT > 16s), bleeding tendency or receiving thrombolytic or anticoagulant therapy;
7. Failed to recover from adverse events (except hair loss) after prior medication use;
8. The patient has any active autoimmune disease or a history of autoimmune disease;
9. Clinical symptoms or diseases of the heart that are not well controlled;
10. Congenital or acquired immune deficiency;
11. Received chemotherapy, targeted and radiotherapy within 2 weeks before enrollment;
12. Concomitant diseases/History:(1) Clinically significant hemoptysis occurred within 3 months before enrollment (hemoptysis > 50ml per day);Or bleeding symptoms of significant clinical significance or a clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occultation and above, or suffering from vasculitis, etc.;(2) Arteriovenous thrombosis events occurred within 6 months before enrollment, such as cerebrovascular accident (including temporary ischemic attack), deep venous thrombosis (except those who had been cured after intravenous catheterization due to chemotherapy) and pulmonary embolism, etc.;(3) hypertension, which cannot be well controlled by antihypertensive drug therapy (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg);During the first 6 months of randomization, myocardial infarction, severe/unstable angina, NYHA grade 2 or higher cardiac dysfunction, clinically significant ventricular arrhythmias or ventricular arrhythmias, and symptomatic congestive heart failure;(4) Interstitial lung disease, non-infectious pneumonia or uncontrollable systemic diseases (e.g., diabetes, pulmonary fibrosis and acute pneumonia);(5) Renal insufficiency: urine protein ≥ ++ indicated by routine urine examination, or confirmed 24-hour urine protein level ≥1.0g; (6) History of live attenuated vaccine vaccination within 28 days prior to initial study administration or expected live attenuated vaccine vaccination during study period;(7) human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS);Active hepatitis (hepatitis B, defined as HBV-DNA ≥ 500 IU/ mL;Hepatitis C, defined as hcV-RNA higher than the lower limit of assay) or co-infection with hepatitis B and c;(8) Severe infection, including but not limited to bacteremia and severe pneumonia requiring hospitalization, occurred within 4 weeks before the first administration;Active infection with CTCAE grade ≥2 requiring systemic antibiotic treatment within 2 weeks prior to initial administration, or fever of unknown origin >38.5°C during screening/prior to initial administration (as determined by the investigator, fever due to tumor can be included);Evidence of active tuberculosis infection within 1 year before administration;(9) Have been diagnosed with any other malignant tumor within 3 years prior to entry into the study;(10) Major surgery performed within 28 days before enrollment (tissue biopsy and peripheral venipuncture placement of central venous catheter [PICC] required for diagnosis are permitted);
13. Subjects who have received or are planning to receive allogeneic bone marrow transplantation or solid organ transplantation;
14. Peripheral neuropathy ≥ grade 2;Patients with active brain metastases, cancerous meningitis, spinal cord compression, or diseases of the brain or pia meningeal found by imaging CT or MRI examination at the time of screening (patients with brain metastases who had completed treatment 14 days before enrollment and had stable symptoms could be enrolled, but were confirmed to have no symptoms of cerebral hemorrhage by craniocerebral MRI, CT or venography evaluation);
15. There are significant factors affecting oral drug absorption, such as inability to swallow, chronic diarrhea, and presence of clinically significant intestinal obstruction.
16. Corrected QT interval > 470 msec;If a patient has a prolonged QT interval, but the investigator assessed the cause of the prolonged QT interval as pacemaker (and no other cardiac abnormalities), discussion with other study physicians will be required to determine whether the patient is eligible for inclusion.
17. Known allergic to pharmaceutical ingredients;
18. Female subjects who are pregnant, breast-feeding, or planning to become pregnant during the study period.
19. Patients with other serious physical or mental disorders or abnormal laboratory tests that may increase the risk of study participation or interfere with study results, and who are considered unsuitable for study participation by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 24 months
  Objective Response Rate

SECONDARY OUTCOMES:
PFS | up to 24 months
  progression-free survival
OS | up to 24 months
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Ruixia Guo, Director, Principal Investigator — The First Affiliated Hospital of Zhengzhou University